CLINICAL TRIAL: NCT03797638
Title: Characterization of Manual Dexterity by Finger Force Manipuladum (FFM) in Patients With Writer's Cramp and in Control Subjects
Acronym: FFM_CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SSA_2018_4
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Dystonic Disorder; Focal Dystonia; Writer's Cramp
Keywords: Dystonic Disorder; Focal Dystonia; Writer's Cramp
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with writer's cramp (Experimental): Patients with writer's cramp
  Interventions: Device: Finger Force Manipuladum (FFM)
- Control subjects (Other): Control subjects, without writer's cramp, matched with case subjects with age, gender and hand writing
  Interventions: Device: Finger Force Manipuladum (FFM)

INTERVENTIONS:
Device: Finger Force Manipuladum (FFM) — Tasks performed with the device Finger Force Manipuladum (FFM), to assess abilities such as finger individuation but also fine finger force control, finger movement regularity and speed.

SUMMARY:
Writer's cramp is a focal dystonia characterized by abnormal movements and postures during writing. Limited finger independence during writing manifests as difficulty suppressing unwanted activations of neighbouring non task-relevant fingers. Patients with Writer's cramp also have difficulty in fine control of grip force.

The investigators have recently developed the Finger Force Manipulandum which quantifies the forces applied by each fingers in different tasks. This method is sensitive for detection and quantification of small unwanted contractions in non-active ('stationary') fingers. Different tasks have been developed to assess abilities such as finger individuation but also fine finger force control, finger movement regularity and speed.

The aim of this study is to assess if developed tasks allow to precisely characterize writer's cramp condition in terms of abilities aforementioned.

To do so, performance of 20 writer's cramp patients in the developed task will be compared with performance of 20 control participants (matched in age, sex and writing hand) in the same tasks.

ELIGIBILITY:
Inclusion criteria for patients with writer's cramp

* Patient with writer's cramp and writing speed <140 letters / min
* Writer's cramp focal dystonia specific to the task of writing
* Patient treated or not with botulinum toxin injection
* Person having attended school in French

Non inclusion criteria for patients with writer's cramp

* Patients whose writer's cramp has no impact on the handwriting and has kept a writing speed> 140 letters per minute.
* Tremor of writing
* Neurological condition other than writer's cramp (eg Parkinson's syndrome)
* Pain, trauma or pathology of the upper limb of the writing member other than the writer's cramp who required medical or surgical treatment in the last 6 months preceding the initial check-up

Inclusion criteria for control subjects

•> 18 years old

* Without writer's cramp
* Person having attended school in French

Non inclusion criteria for control subjects

* Tremor of writing
* Neurological condition other than writer's cramp (eg Parkinson's syndrome)
* Pain, trauma or pathology of the upper limb of the writing member other than the writer's cramp who required medical or surgical treatment in the last 6 months preceding the initial check-up

Matching criteria between cases and control patients

* Age (± 5 years)
* Gender
* Hand writing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Manual dexterity by the FFM | Inclusion
  Compare the manual dexterity by the FFM between subjects with writer's cramp and control subject

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BLETON, PhD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided